CLINICAL TRIAL: NCT01364168
Title: Prospective Cohort With Incident Stroke
Acronym: PROSCIS
Status: Recruiting | Type: Observational
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Martin Dichgans, Prof., Ludwig-Maximilians - University of Munich
Other Study IDs: ISD-PROSCIS-01
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- First ever acute ischemic stroke: Patients over 18 years and without prior stroke according to WHO criteria, displaying an ischemic stroke, onset within the last 7 days, language German

SUMMARY:
The primary aim of the study is to derive and validate risk scores for vascular endpoints (recurrent stroke, myocardial infarction, and other complications of stroke) and for death following an incident stroke. For this purpose patients with an incident stroke will be followed for 36 months with additional assessments at 3, 12, 24 and 36 months.

DETAILED DESCRIPTION:
Risk of vascular disease including stroke, myocardial infarction, and vascular death is high after stroke but there are only few prognostic models for long term risk up to 3 years. About 850 patients with an incident stroke will be followed for 3 years with assessments at baseline and at 3, 12, 24, and 36 months. Factors that have already been reported to be significant predictors of vascular diseases in previous studies as well as new biomarkers (e.g. neuroimaging, blood based biomarkers) identified in this cohort will be considered. The improvement of discrimination including these new variables in the models will be investigated. Several measures of improving predictive properties (e.g. calibration, discrimination, net reclassification) will be used to compare predictive models with different complexity. The model will be validated using the bootstrap method (internal validation) and an independent external sample in cooperation with the prospective CSB-stroke cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Language: German
* First ever acute ischemic stroke that occurred with stroke onset in the last 7 days
* Written informed consent by patient prior to study participation
* Willingness to participate in follow-up

Exclusion Criteria:

* Prior stroke (definition according to WHO criteria)
* Patients presenting brain tumour or brain metastasis
* Participation in an intervention- / AMG-study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to a specialized stroke service because of an acute stroke
Sampling Method: Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2011-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Combined vascular endpoint composed of stroke, myocardial infarction, and vascular death | 36 months
  This evaluation will be based on a structured interview with the patient. In case of positive screening more information will be obtained by hospital or physician.

SECONDARY OUTCOMES:
Combined vascular endpoint composed of stroke, myocardial infarction, and vascular death | 24 months
  This evaluation will be based on a structured interview with the patient. In case of positive screening more information will be obtained by hospital or physician. In case of death of the patient, evaluation will be based on data from the registry office.
Combined vascular endpoint composed of stroke, myocardial infarction, and vascular death | 12 months
  This evaluation will be based on a structured interview with the patient. In case of positive screening more information will be obtained by the physician. In case of death of the patient, evaluation will be based on data from the registry office.
Course of cognitive function | 36 months
  This evaluation will be based on a structured interview with the patient. In case of positive screening more information will be obtained by the physician.
Course of depression | 36 months
  This evaluation will be based on a structured interview with the patient. In case of positive screening more information will be obtained by the physician.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dichgans, Prof., Study Chair — Institute for Stroke and Dementia Research, Klinikum der Universität München
Locations (2):
- Germany (2):
  - Center for Stroke Research Berlin, Charité Universitätsmedizin Berlin, Berlin
  - Interdisciplinary Stroke Center Munich, Klinikum der Universität München, Munich

REFERENCES:
- [Background] Liman TG, Zietemann V, Wiedmann S, Jungehuelsing GJ, Endres M, Wollenweber FA, Wellwood I, Dichgans M, Heuschmann PU. Prediction of vascular risk after stroke - protocol and pilot data of the Prospective Cohort with Incident Stroke (PROSCIS). Int J Stroke. 2013 Aug;8(6):484-90. doi: 10.1111/j.1747-4949.2012.00871.x. Epub 2012 Aug 29. PMID 22928669
- [Result] Malsch C, Liman T, Wiedmann S, Siegerink B, Georgakis MK, Tiedt S, Endres M, Heuschmann PU. Outcome after stroke attributable to baseline factors-The PROSpective Cohort with Incident Stroke (PROSCIS). PLoS One. 2018 Sep 26;13(9):e0204285. doi: 10.1371/journal.pone.0204285. eCollection 2018. PMID 30256828
- See also: Related Info — http://www.klinikum.uni-muenchen.de/Institut-fuer-Schlaganfall-und-Demenzforschung/de/index.html
- See also: Related Info — http://www.klinikum.uni-muenchen.de/Interdisziplinaeres-Schlaganfallzentrum/en/index.html